CLINICAL TRIAL: NCT00827762
Title: Behavioral Effects of Kuvan in Children With Mild Phenylketonuria
Status: Terminated | Type: Observational
Why Stopped: Too few participants recruited within timeframe
Sponsor: Washington University School of Medicine (Other)
Collaborators: BioMarin Pharmaceutical (Industry); University of Missouri-Columbia (Other); Northwestern University (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: MildPKU/Kuvan/White
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Phenylketonuria
Keywords: phenylketonuria; Kuvan; sapropterin; behavior; cognition; executive abilities; attention
MeSH Terms: conditions — Phenylketonurias; Behavior | interventions — sapropterin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Phenylketonuria: Individuals with mild phenylketonuria/hyperphenylalanemia who are beginning treatment with Kuvan.
  Interventions: Drug: Kuvan

INTERVENTIONS:
Drug: Kuvan — 20/mg/kg/day taken once daily or as otherwise prescribed by physician as standard care.
  Other Names: Sapropterin

SUMMARY:
The purpose of this study is to determine whether improvements in behavior occur in children with phenylketonuria (PKU) who are taking Kuvan.

DETAILED DESCRIPTION:
Little research has been conducted to examine behavior and cognition in children with mild PKU/hyperphenylalanemia, but there is evidence of reductions in general intelligence (IQ) (Costello, 1994) and impairments in executive abilities (Diamond, 1994; Gassio, 2005) in this population. It is important to note that the phenylalanine levels of children with mild PKU are approximately equivalent to those of children with classical PKU whose phenylalanine levels have been managed through dietary control. In children with diet-treated PKU, impairments in behavior and cognition are well-documented, particularly in relation to executive abilities (Christ, 2006; White, 2001, 2002). Taken together, these findings suggest that children with mild PKU are at risk for behavioral and cognitive impairments, and it is possible that these impairments may be mitigated by lowering phenylalanine levels through treatment with Kuvan.

To investigate this issue, approximately 20 children with mild PKU from 6 to 18 years of age (inclusive) and their parents will participate in the study. The behavior and cognition of children with mild PKU will be assessed using the following methods: (1) Parents will complete inventories to rate the behavior and cognition of their children; (2) Older children will complete self-report inventories to rate their behavior and cognition; (3) Cognitive tasks assessing IQ and executive aspects of attention (i.e., sustained attention and inhibitory control) will be administered to all children.

The primary objectives are two-fold. First, we will determine if behavior and cognition are compromised in children with mild PKU prior to treatment with Kuvan (baseline). To accomplish this objective, we will administer measures of behavior and cognition that include normative data based on age. We hypothesize that children with mild PKU will have ratings and scores that are ≥ 1 standard deviation from the normative mean. Second, we will determine if behavior and cognition improve in children with mild PKU following treatment with Kuvan. To accomplish this objective, we will administer the same measures of behavior and cognition after 4 and 24 weeks of treatment with Kuvan(4-week and 24-week follow-ups, respectively). We hypothesize that the follow-up ratings and scores of children with mild PKU will improve by ≥ 0.5 standard deviation relative to their baseline ratings and scores.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and/or assent.
* Willing and able to comply with study procedures.
* Between 6 and 18 years of age, inclusive.
* Intention of physician to prescribe Kuvan.
* Phenylalanine levels between 360μmol/L and 600μmol/L, inclusive, when untreated with dietary restrictions.
* Negative pregnancy test if of childbearing potential.
* Willing to use contraception if sexually active.

Exclusion Criteria:

* Treatment with Kuvan within the past 6 months.
* Pregnant, breastfeeding, or planning to become pregnant during study.
* Use of investigational product less than 30 days prior to or during study.
* Concurrent condition that could interfere with participation or safety.
* Any condition creating high risk of poor compliance with study.
* History of major medical disorder unrelated to phenylketonuria.
* Perceived to be unreliable or unavailable for study.
* Use of L-Dopa, methotrexate, or other drugs that inhibit folate metabolism.
* Known hypersensitivity to sapropterin or excipients.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care clinic for phenylketonuria.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) | baseline, 4-week follow-up, 24-week follow-up

SECONDARY OUTCOMES:
Behavior Assessment System for Children - Second Edition (BASC-2) | baseline, 4-week follow-up, 24-week follow-up
Conners 3rd Edition (Conners 3) | baseline, 4-week follow-up, 24-week follow-up
Conners Continuous Performance Test II Version 5 (CCPT-II Version 5) | baseline, 4-week follow-up, 24-week follow-up
Matrix Reasoning subtest of the Wechsler Abbreviated Scale of Intelligence (WASI) | baseline, 4-week follow-up, 24-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Desiree White, Ph.D., Principal Investigator — Washington University School of Medicine; Dorothy K. Grange, M.D., Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Northwestern University/Children's Memorial Hospital, Chicago, Illinois
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Background] Christ SE, Steiner RD, Grange DK, Abrams RA, White DA. Inhibitory control in children with phenylketonuria. Dev Neuropsychol. 2006;30(3):845-64. doi: 10.1207/s15326942dn3003_5. PMID 17083296
- [Background] White DA, Nortz MJ, Mandernach T, Huntington K, Steiner RD. Age-related working memory impairments in children with prefrontal dysfunction associated with phenylketonuria. J Int Neuropsychol Soc. 2002 Jan;8(1):1-11. PMID 11843066
- [Background] White DA, Nortz MJ, Mandernach T, Huntington K, Steiner RD. Deficits in memory strategy use related to prefrontal dysfunction during early development: evidence from children with phenylketonuria. Neuropsychology. 2001 Apr;15(2):221-9. doi: 10.1037//0894-4105.15.2.221. PMID 11324865